CLINICAL TRIAL: NCT01138488
Title: A Trial Investigating the Pharmacokinetic Properties of NN5401 in Children, Adolescents and Adults With Type 1 Diabetes
Brief Title: A Trial Investigating the Total Exposure of NN5401 (Insulin Degludec/Insulin Aspart) in Children, Adolescents and Adult Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Collaborators: HNEC TEST (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-1982; U1111-1113-6874 (Other: WHO); 2009-016779-31 (EudraCT Number)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NN5401 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Insulin degludec/insulin aspart administered as a single subcutaneous injection (under the skin).

SUMMARY:
This trial was conducted in Europe. The aim of this study was to investigate the total exposure of NN5401 (insulin degludec/insulin aspart) in children, adolescents and adult subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index for children: 15.0-20.0 kg/m^2 (both inclusive), for adolescents: 18.0-28.0 kg/m^2 (both inclusive) and for adults maximum 30.0 kg/m^2

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month, or more than 500 mL within 3 months prior to screening
* Not able or willing to refrain from smoking during the inpatient period
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration-time curve | from 0 to infinity after single-dose
Area under the serum insulin aspart concentration-time curve | from 0 to 12 hours after single-dose

SECONDARY OUTCOMES:
Maximum observed insulin degludec concentration of NN5401 (insulin degludec/insulin aspart) observed | from 0 to 57 hours after single-dose
Maximum observed insulin aspart concentration of NN5401 (insulin degludec/insulin aspart) observed | from 0 to 12 hours after single-dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hanover, Germany

REFERENCES:
- [Result] Biester T, Danne T, Blasig S, Remus K, Aschemeier B, Kordonouri O, Bardtrum L, Haahr H. Pharmacokinetic and prandial pharmacodynamic properties of insulin degludec/insulin aspart in children, adolescents, and adults with type 1 diabetes. Pediatr Diabetes. 2016 Dec;17(8):642-649. doi: 10.1111/pedi.12358. Epub 2016 Jan 18. PMID 26782928
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com